CLINICAL TRIAL: NCT07024654
Title: A Prospective Case Series: Genicular Embolization Using Doxycycline Sclerotherapy
Brief Title: Genicular Embolization Using Doxycycline Sclerotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Campbell Clinic (Other)
Responsible Party: Principal Investigator, Joshua Brandon, Principal Investigator, Campbell Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-10650-FB
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Chronic Knee Pain; Osteoarthritis
Keywords: Chronic knee pain; osteoarthritis; genicular sclerotherapy
MeSH Terms: conditions — Osteoarthritis | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: single-group, prospective interventional pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Doxycycline Genicular Sclerotherapy Arm (Experimental): Participants in this arm will undergo sclerotherapy using doxycycline to target terminal genicular arteries associated with knee pain. The procedure is performed under ultrasound guidance, and the goal is to evaluate the safety and potential efficacy of doxycycline as a sclerosing agent for managing chronic knee pain symptoms.
  Interventions: Drug: Doxycycline Injection

INTERVENTIONS:
Drug: Doxycycline Injection — Injection of doxycycline as a sclerosing agent into the genicular artery region under ultrasound guidance for the purpose of evaluating its effectiveness in reducing knee pain.
  Other Names: Ultrasound Guided Sclerotherapy

SUMMARY:
The goal of this prospective case series is to develop an alternative pain management procedure for patients who are not surgical candidates. The main question it aims to answer is: Is genicular sclerotherapy using doxycycline a safe and effective pain management option for patients with chronic knee pain who are not surgical candidates?

OUTCOME MEASURES:

Primary: Visual Analog Scale (VAS) score at 3 months

Secondary:

* VAS at 12 months
* Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score at 12 months

DETAILED DESCRIPTION:
The purpose of this study is to develop an alternative pain management procedure for patients who are not surgical candidates. Using sclerotherapy (a procedure in which a medication is injected into small blood vessels causing them to scar, shrink and collapse) in the small terminal branches of some of the blood vessels in the knee, the aim is to adapt this proven therapy for varicose veins, cysts, and vascular malformations to pain management. Doxycycline will be used as the injectable to perform the procedure. Doxycyline is a FDA approved medication commonly used for bacterial infections and is is frequently used off-label as a sclerosing agent; however, it is not specifically FDA approved for use in sclerotherapy.

This is a pilot study. A pilot study is a small-scale, preliminary study conducted before a larger, more comprehensive research project. Its purpose is to test and refine the research methods, procedures, and instruments, ensuring they are feasible, practical, and reliable.

Visit 1: Consent and treatment procedure: Subjects will be consented and baseline VAS (visual analog scale) and WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index)will be obtained. Procedure will be performed by one of the study providers as follows: Following sterile cleaning of the skin and administration of lidocaine to anesthetize injection tract, ultrasound guidance will be utilized to isolate target sites of the peripheral vasculature of the genicular artery in one knee. Up to four sites in the index knee may be injected as needed based on pain presentation and physician's discretion. A maximum of 100 milligrams of doxycycline diluted in 10 milliliters of sterile water will be used per subject. Post procedure icing will be performed for 15 minutes to help prevent the occurrence of ischemia and bruising.

Post-operatively, a prescription for either Lortab or Tramadol will be offered and an over the counter pain medication option will be recommended.

If the subject experiences an adverse event, please contact the study provider for an exam, lab-work and/or consultation as needed.

Following the procedure, restrict activity for 1-2 weeks to protected weight bearing and to advance as tolerated.

Visit 2: 2 weeks post-op: Follow up appointment in clinic with provider. VAS and WOMAC will be collected. Any problems/concerns the patient may be having and if the subject is considering seeking other treatment will be discussed and documented.

Visit 3: 6 weeks post-op: Follow up appointment in clinic with provider. VAS and WOMAC will be collected. Any problems/concerns the patient may be having and if the subject is considering seeking other treatment will be discussed and documented.

Visit 4: 3 months post-op: Follow up appointment in clinic with provider. VAS and WOMAC will be collected. Any problems/concerns the patient may be having and if the subject is considering seeking other treatment will be discussed and documented.

Visit 5: 6 months post-op: VAS and WOMAC will be collected over the phone. Any problems/concerns the patient may be having and if the subject is considering seeking other treatment will be discussed and documented.

Visit 6: 9 months post-op: VAS and WOMAC will be collected over the phone. Any problems/concerns the patient may be having and if the subject is considering seeking other treatment will be discussed and documented.

Visit 7: 12 months post-op: VAS and WOMAC will be collected over the phone. Any problems/concerns the patient may be having and if the subject is considering seeking other treatment will be discussed and documented.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age or older.
* KL Score 2-3
* VA Grade >5
* Native knee
* Willing and able to provide consent.
* Willing and able to complete questionnaires.
* Willing and able to complete follow up visits.
* Speak and write fluent English
* Unilateral knee (if bilateral knee pain, identify knee for procedure)
* All subjects may be included regardless of sex. Women must be either surgically sterilized postmenopausal defined as having no menstrual periods for 12 consecutive months

Exclusion Criteria:

* Allergies to doxycycline or any other substances used in procedure
* Steroid injection in the index knee within the last 90 days
* Knee surgery on index knee in the last 180 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 3 months post-op
  Primary outcome measure will be visual analog scale scores at 3 months post-op. Scores 0-10, 0 being no pain, 10 being the worst pain.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 1 year post-op
  Secondary outcome measure will be Western Ontario and McMaster Universities Osteoarthritis Index scores at 1 year.
  Scores scale from 0 (no symptoms) to 96 (maximum pain, stiffness, and physical dysfunction)
Visual Analog Scale (VAS) | 1 year post-op
  Secondary outcome measure will be visual analog scale scores at 1 year post-op. Scores 0-10, 0 being no pain, 10 being the worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Brandon, MD, Principal Investigator — Campbell Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bountouroglou DG, Azzam M, Kakkos SK, Pathmarajah M, Young P, Geroulakos G. Ultrasound-guided foam sclerotherapy combined with sapheno-femoral ligation compared to surgical treatment of varicose veins: early results of a randomised controlled trial. Eur J Vasc Endovasc Surg. 2006 Jan;31(1):93-100. doi: 10.1016/j.ejvs.2005.08.024. Epub 2005 Oct 17. PMID 16233981
- [Background] Wong MN, Murakami JW. Doxycycline Sclerotherapy of Mandibular Aneurysmal Bone Cysts: A Brief Clinical Study. J Craniofac Surg. 2025 Jan-Feb 01;36(1):e31-e33. doi: 10.1097/SCS.0000000000010697. Epub 2024 Sep 23. PMID 39311568
- [Background] McDermott D, Wakefield D, Kowalsky M, Sethi P, Vitale MA, Morrey BF. Intrabursal Doxycycline Sclerotherapy for Recurrent Olecranon Bursitis of the Elbow: A Case Control Study. J Hand Surg Glob Online. 2024 Apr 8;6(4):504-509. doi: 10.1016/j.jhsg.2024.03.006. eCollection 2024 Jul. PMID 39166200
- [Background] Liu S, Swilling D, Morris EM, Macaulay W, Golzarian J, Hickey R, Taslakian B. Genicular Artery Embolization: A Review of Essential Anatomic Considerations. J Vasc Interv Radiol. 2024 Apr;35(4):487-496.e6. doi: 10.1016/j.jvir.2023.12.010. Epub 2023 Dec 19. PMID 38128722
- [Background] Torkian P, Golzarian J, Chalian M, Clayton A, Rahimi-Dehgolan S, Tabibian E, Talaie R. Osteoarthritis-Related Knee Pain Treated With Genicular Artery Embolization: A Systematic Review and Meta-analysis. Orthop J Sports Med. 2021 Jul 14;9(7):23259671211021356. doi: 10.1177/23259671211021356. eCollection 2021 Jul. PMID 34350303
- [Background] van Zadelhoff TA, Moelker A, Bierma-Zeinstra SMA, Bos PK, Krestin GP, Oei EHG. Genicular artery embolization as a novel treatment for mild to moderate knee osteoarthritis: protocol design of a randomized sham-controlled clinical trial. Trials. 2022 Jan 8;23(1):24. doi: 10.1186/s13063-021-05942-x. PMID 34998425